CLINICAL TRIAL: NCT03662230
Title: Incidence and Severity of Acute Respiratory Distress Syndrome (ARDS) in the French Wounded Soldiers
Acronym: SDRA-OPEX
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: SDRA-OPEX
Record Dates: First submitted 2018-07-23; First posted 2018-09-07 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2019-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: war wounds; intensive care unit
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the incidence of the ARDS in the French wounded soldiers.

DETAILED DESCRIPTION:
The Acute Respiratory Distress Syndrome (ARDS) complicates war wounds. Among the repatriated wounded persons, it can appear in the first 7 days.

It has been well described among American soldiers and it is known that it's serious, frequent and multifactorial.

However, not a single study has described the frequency and the severity of the ARDS in French wounded soldiers.

Thus the purpose of this study is to estimate the incidence and severity of the ARDS among the French wounded soldiers, admitted in continuing care and intensive care unit between 2001 and 2017.

The analysis of this data collection will let us improve the medical care of the ARDS in Outside Operation.

ELIGIBILITY:
Inclusion Criteria:

* Patient evacuated from the theatre of outside operation and hospitalized in intensive care unit in France between 2001 et 2017

Exclusion Criteria:

* Opposition to the use of personal data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient evacuated from the theatre of outside operation and hospitalized in intensive care unit in France between 2001 et 2017
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of ARDS | Day 7
  The appearance of ARDS is defined by a ratio of partial pressure arterial oxygen (PaO2) and fraction of inspired oxygen (FiO2) lower than 300 in 7 days after the wound.

SECONDARY OUTCOMES:
Assess the severity of ARDS | 7 days
  the severity of ARDS will be assessed regarding the necessity or not of non-invasive and invasive ventilation
Description of the severity of ARDS | 7 days
  the therapeutic intensity will be describe with : Maximal Positive end-expiration pressure (PEEP), curarisation, nitrogen monoxide (NO), prone position , Extracorporeal membrane oxygenation.
Mortality | Day 90
  Assess the mortality since hospitalization
Assessment of the severity of ARDS | 7 days
  the severity of ARDS will be assessed regarding duration of non-invasive and invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Julien Bordes, professor, Study Director — Hopital d'Instruction des Armées Sainte Anne
Locations (1):
- Hôpital d'Instruction des Armées Sainte Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No